CLINICAL TRIAL: NCT05857553
Title: Unconditional Cash Transfers to Address Poverty as a Fundamental Cause of Child Welfare Involvement
Brief Title: Cash Transfers to Address Child Welfare Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Redlich Horwitz Foundation (Unknown); Rutgers University (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Stacia West, Associate Professor & Co-Founding Director of the Center for Guaranteed Income Research, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OCFS DCT Pilot
Record Dates: First submitted 2023-04-28; First posted 2023-05-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Child Poverty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in the treatment group will receive $500 per month for 12 months
  Interventions: Other: Unconditional Cash Transfer
- Control Group (Active Comparator): Participants in the control group will not receive monthly cash benefits.
  Interventions: Other: No Direct Cash Transfer

INTERVENTIONS:
Other: Unconditional Cash Transfer — Unconditional monthly transfer of $500 to household
  Other Names: Direct Cash Transfer; Guaranteed Income
  Arms: Treatment Group
Other: No Direct Cash Transfer — No intervention
  Arms: Control Group

SUMMARY:
In partnership with New York Office of Child and Family Services (OCFS), investigators will execute a randomized controlled trial to determine the impacts of unconditional cash transfers of $500 per month for 12 months. Investigators will measure the impacts of the unconditional cash transfers on parental physical and mental health, child health and healthcare utilization, financial stability, and interactions with the child welfare system.

DETAILED DESCRIPTION:
Poverty has been identified as a powerful predictor of child maltreatment and child welfare involvement. Recent research shows that even modest economic and concrete supports are associated with reduced child maltreatment and involvement with child welfare. Toward that end, the New York State Office of Children and Family Services (OCFS), in partnership with the Office of Temporary Disability Assistance (OTDA) and the Center for Guaranteed Income Research (CGIR), University of Pennsylvania is conducting on randomized controlled trial of unconditional cash transfers among families with prior child welfare referrals in three New York counties in 2023.

The project will enroll approximately 150 households in Monroe, Onondaga, and Westchester counties to receive $500 per month, unconditionally, over a one-year period, totaling $6,000 per family. Another 300 will be assigned to the control group and will not receive the unconditional cash transfers but will be eligible to participate in research activities. Families will be eligible if they were served through differential response, called Family Assessment Response (FAR) in New York State. FAR is used for CPS reports that have been accepted by the New York State Central Register for Child Abuse and Maltreatment (SCR) where there is no safety concern that rises to the level of immediate or impending danger for the child and/or family. Often, families served in the FAR track have been referred for poverty-related social needs.

Randomized Controlled Trial Design: Households referred and determined eligible for Family Assessment Response (FAR) will be invited to participate in a randomized controlled trial of unconditional cash transfers. Approximately 150 individuals will be randomly assigned to the treatment group and will receive the $500 unconditional cash transfers for one year. Another 300 will be assigned to the control group and will not receive the unconditional cash transfers but will be eligible to participate in research activities. Youth Research Inc. (YRI), an agency contracted by the New York Office of Child and Family Services (OCFS), will disburse funds on a debit card. me but will be invited to participate in compensated research activities. Longitudinal repeated measures will be utilized through surveys conducted at baseline, 6 months, 12 months, and 18 months. Future involvement with child welfare will be measured using linked administrative data from OCFS.

ELIGIBILITY:
To participate in this pilot, caregivers must meet the following eligibility criteria:

* Received an invitation from an OCFS caseworker to apply
* Have met the state eligibility requirements for the Family Assessment Response (FAR) within the previous six months
* Live in Monroe, Onondaga, or Westchester County, New York
* Be 18 years of age or older at the time of application.

Exclusion criteria:

● Self-reported enrollment in another cash transfer study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Unfounded reports to CPS | 18 months
  Count of unfounded reports using CPS administrative data
Investigative Track reports to CPS | 18 months
  Count of Investigative Track using CPS administrative data
Indicated reports to CPS | 18 Months
  Count of Indicated reports using CPS administrative data
Substantiated reports to CPS | 18 Months
  Count of Substantiated reports using CPS administrative data
Family Assessment Response (FAR) track reports to CPS | 18 months
  Count of Family Assessment Response (FAR) track reports using CPS administrative dat
Unsubstantiated reports to CPS | 18 months
  Count of Unsubstantiated reports using CPS administrative data
Foster care placements | 18 months
  Count of Foster care placements using CPS administrative data

SECONDARY OUTCOMES:
Parental self-reported general health (SF-36) | 12 months
  Average of 5-point likert scale score on 5 questions
Mental health (Kessler 10) | 12 months
  Each item is scored from one 'none of the time' to five 'all of the time'. Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
Stress and coping (Perceived Stress Scale - 4) | 12 months
  Each item is scored from "never" to "all of the time" on a 5-point scale. Scores of 4 items are then summed, yielding a minimum score of 0 and a highest score of 16. Higher scores are correlated to more stress
Family dynamics and parenting (CHAOS) | 12 months
  Each item is scored "yes" or "no". Scores of the items are then summed. The higher the score the higher the level of environmental chaos in the home.
Parental Stress Sale | 12 months
  18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). Each item is scored on a 5-point Likert scale. Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Food insecurity | 12 months
  Answer to single item question "In the past four weeks, did you worry that your household would not have enough food?"
Child missed medical care | 12 months
  Parental yes/no report of any child in home with missed medical care in preceding 6 months
Child school truancy | 12 months
  Parental report of day of missed school for each child in the home aged 6-17 in the preceding 6 months
Hours per week of relative childcare | 12 months
  Parent-reported number of hours each week each child 0-5 spends receiving care from a relative other than a parent or guardian
Hours per week of non-relative childcare | 12 hours
  Parent-reported number of hours each week each child 0-5 spends receiving care from a non-relative
Hours per week of formal childcare | 12 months
  Parent-reported number of hours each week each child 0-5 spends receiving care in a day care center, preschool, or prekindergarten
Financial-well being (CFPB Financial Well-Being Scale | 12 months
  Each item is scored 0 to 4 and summed to a total. The sum total is then converted to a total response value on the CFPB Financial Well-Being Scale score from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Stacia West, PhD, Principal Investigator — University of Pennsylvania/University of Tennessee
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05857553/Prot_SAP_000.pdf